CLINICAL TRIAL: NCT03191591
Title: The First 1,000 Days Program: Maternal-Child Obesity Prevention in Early Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Boston Foundation (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Elsie Taveras, MD, Chief, Division of General Academic Pediatrics, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016P000801; 1K24DK105989 (NIH)
Record Dates: First submitted 2017-06-09; First posted 2017-06-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Overweight and Obesity; Social Determinants of Health; Physical Activity; Sleep; Feeding Behavior; Diet Habit
Keywords: Overweight; Obesity; Maternal-child; Social Determinants of Health
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The First 1,000 Days program is a systems-level program that will reach all expectant mothers and families with 0-2 year olds receiving care at Boston-area community health centers. Mothers and infants at two similar non-intervention Boston-area health centers will be used as a comparison sample. Maternal and infant obesity-related clinical information is routinely recorded during patient visits in the EHR used at both the intervention and comparison sites. Sample size enrollment reflects maternal-infant dyads.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First 1,000 Days Program (Experimental)
  Interventions: Behavioral: First 1,000 Days Program Site

INTERVENTIONS:
Behavioral: First 1,000 Days Program Site — Program components will include 1) Enhancements to and improved use of electronic health records to improve the quality of preventive services and screening for social determinants of health; 2) Staff and provider training; 3) Consistent behavior change messaging; 4) Patient education via print materials, text messaging and short videos; and 5) Strengthening the integration of clinical and public health services to support behavior change and address social determinants of health.

SUMMARY:
The First 1000 Days (conception to age 2) is a crucial period for the development and prevention of obesity and its adverse consequences in mother-child pairs and their families. The overall aim of the First 1000 Days program is to work across early-life systems to prevent obesity, promote healthy routines and behaviors, address social determinants of health, and reduce health disparities among vulnerable children and families at community health centers in the Boston, MA area.

The study aims to simultaneously implement and evaluate an obesity prevention program across early life systems to reduce the prevalence of obesity risk factors within racial/ethnic minority families, close the gap in maternal-child health disparities, and assess and address social determinants of health.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women receiving prenatal care at select community health centers in the Boston, MA area
* All families of children aged 0-2 years receiving pediatric care at select community health centers in the Boston, MA area

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1645 (Estimated)
Dates: Start 2016-08-09 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Maternal Gestational Weight Gain | First prenatal care visit to 36 weeks gestation
  Weight gained during pregnancy
Infant Weight-for-Length Z-Score | Child age 6 months
  Age- and sex-specific weight-for-length z-score
Infant Weight-for-Length Z-score | Child age 12 months
  Age- and sex-specific weight-for-length z-score
Infant Weight-for-Length Z-Score | Child age 24 months
  Age- and sex-specific weight-for-length z-score

SECONDARY OUTCOMES:
Change from 1st trimester maternal diet to 3rd trimester | An average of 18 weeks (1st trimester to 3rd trimester)
  Average weekly intake
Change from 1st trimester maternal physical activity to 3rd trimester | An average of 18 weeks (1st trimester to 3rd trimester)
  Days per week physically active for at least 30 minutes per day
Change from 1st trimester maternal sleep duration to 3rd trimester | An average of 18 weeks (1st trimester to 3rd trimester)
  Average hours per day
Change from 1st trimester maternal sedentary time to 3rd trimester | An average of 18 weeks (1st trimester to 3rd trimester)
  Hours per day of screentime
Change from 1st trimester depression to 3rd trimester | An average of 18 weeks (1st trimester to 3rd trimester)
  Edinburgh Postnatal Depression Scale
Change from 1st trimester maternal food insecurity to 3rd trimester | An average of 18 weeks (1st trimester to 3rd trimester)
  2-question validated scale
Change from 1st trimester maternal housing insecurity to 3rd trimester | An average of 18 weeks (1st trimester to 3rd trimester)
  2-question validated scale
Change from 1st trimester pregnancy-related anxiety to 3rd trimester | An average of 18 weeks (1st trimester to 3rd trimester)
  5-question validated scale
Change from 1st trimester enrollment in food assistance programs to 3rd trimester | An average of 18 weeks (1st trimester to 3rd trimester)
  Yes/No response options for program enrollment in WIC and SNAP

CONTACTS AND LOCATIONS:
Overall Officials: Elsie Taveras, MD, MPH, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neri Mini F, Saltzman JA, Simione M, Luo M, Perkins ME, Roche B, Blake-Lamb T, Kotelchuck M, Arauz-Boudreau A, Davison K, Taveras EM. Expectant Fathers' Social Determinants of Health in Early Pregnancy. Glob Pediatr Health. 2020 Nov 27;7:2333794X20975628. doi: 10.1177/2333794X20975628. eCollection 2020. PMID 33294495
- [Background] Cheng ER, Luo M, Perkins M, Blake-Lamb T, Kotelchuck M, Arauz Boudreau A, Taveras EM. Household food insecurity is associated with obesogenic health behaviours among a low-income cohort of pregnant women in Boston, MA. Public Health Nutr. 2023 May;26(5):943-951. doi: 10.1017/S1368980022000714. Epub 2022 Mar 24. PMID 35321774
- [Background] Cruz-Bendezu AM, Lovell GV, Roche B, Perkins M, Blake-Lamb TL, Taveras EM, Simione M. Psychosocial status and prenatal care of unintended pregnancies among low-income women. BMC Pregnancy Childbirth. 2020 Oct 12;20(1):615. doi: 10.1186/s12884-020-03302-2. PMID 33046003
- [Background] Blake-Lamb T, Boudreau AA, Matathia S, Tiburcio E, Perkins ME, Roche B, Kotelchuck M, Shtasel D, Price SN, Taveras EM. Strengthening integration of clinical and public health systems to prevent maternal-child obesity in the First 1,000Days: A Collective Impact approach. Contemp Clin Trials. 2018 Feb;65:46-52. doi: 10.1016/j.cct.2017.12.001. Epub 2017 Dec 7. PMID 29225195
- [Background] Simione M, Moreno-Galarraga L, Perkins M, Price SN, Luo M, Kotelchuck M, Blake-Lamb TL, Taveras EM. Effects of the First 1000 Days Program, a systems-change intervention, on obesity risk factors during pregnancy. BMC Pregnancy Childbirth. 2021 Oct 27;21(1):729. doi: 10.1186/s12884-021-04210-9. PMID 34706698
- [Result] Blake-Lamb T, Boudreau AA, Matathia S, Perkins ME, Roche B, Cheng ER, Kotelchuck M, Shtasel D, Taveras EM. Association of the First 1,000 Days Systems-Change Intervention on Maternal Gestational Weight Gain. Obstet Gynecol. 2020 May;135(5):1047-1057. doi: 10.1097/AOG.0000000000003752. PMID 32282612
- [Result] Taveras EM, Perkins ME, Boudreau AA, Blake-Lamb T, Matathia S, Kotelchuck M, Luo M, Price SN, Roche B, Cheng ER. Twelve-Month Outcomes of the First 1000 Days Program on Infant Weight Status. Pediatrics. 2021 Aug;148(2):e2020046706. doi: 10.1542/peds.2020-046706. PMID 34326179